CLINICAL TRIAL: NCT06039410
Title: ISO-101 a Novel Device for the Treatment of Orthostatic Hypotension - a Signal of Efficacy Study
Brief Title: A Novel Device for the Treatment of Postural Hypotension - a Signal of Effectiveness Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isotech Ltd (Industry)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISO0001
Record Dates: First submitted 2023-09-01; First posted 2023-09-15 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Intervention Model Description: Thus, the study is a single centre, unblinded, pre-post study. All participants will act as their own control, and all will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): ISO-101 Device
  Interventions: Device: ISO-101

INTERVENTIONS:
Device: ISO-101 — ISO-101 is an experimental wearable class 1 medical device which when used is able to raise the blood pressure upon standing via controlled isometric muscular contractions

SUMMARY:
The goal of this clinical trial is to test a novel medical device (ISO-101) in patients diagnosied with orthostatic hypotension. The main question[s] it aims to answer are:

* to determine whether the ISO-101 device demonstrates a signal of efficacy in people with OH and whether it is worthy of further clinical evaluation.
* Assess the safety and performance of the ISO-101 device in patients with orthostatic hypotension.

Participants will use the device under controlled conditions and have the following parameters measured before and after standing up:

* blood pressure
* markers of peripheal vascular resistence
* sympathetic nervous system activity measure before and after standing up

DETAILED DESCRIPTION:
This is a proof of principle study aimed at evaluating if there is a signal of efficacy from use of the ISO-101 device in people with orthostatic hypotension. The study is a single centre, unblinded, pre-post study. All participants will act as their own control, and all will receive the intervention.The primary objective is to determine whether the ISO-101 device demonstrates a signal of efficacy in people with OH and whether it is worthy of further clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Adults aged over 18 years with a clinical diagnosis of orthostatic hypotension
* A drop in systolic BP of ≥20 mmHg (with or without a drop in diastolic BP ≥10 mmHg) within 3 minutes of standing up from a supine position
* Able to stand up from a supine position (with assistance if required)

Exclusion Criteria:

* Cognitively unable to follow research procedures
* Physically unable to use the ISO-101 device (e.g., unilateral arm weakness due to stroke)
* Acute or reversible cause of OH (e.g., haemorrhage or sepsis)
* Current pregnancy
* Participants on insulin (participants will be asked to refrain from breakfast on the morning of their assessment)
* Resting supine systolic BP ≥180 or diastolic ≥110 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (mmHg) | From date of enrollment until end of study completion (24 hours)
  The change in resting BP, standing BP and postural BP drop during and immediately after using the device.
Adverse Events | From date of enrollment until end of study completion (24 hours)
  Adverse events

SECONDARY OUTCOMES:
Blood pressure | From date of enrollment until end of study completion (24 hours)
  Magnitude and duration of treatment effect on blood pressure
Cardiovascular variablity | From date of enrollment until end of study completion (24 hours)
  Changes in peripheral vascular resistance (dyn*s*m2/cm5) and sympathetic nervous system activity (heart rate variability)
Erganomics | From date of enrollment until end of study completion (24 hours)
  Number of participants able to effectively use the device
Post study participant questionaire | From date of enrollment until end of study completion (24 hours)
  7 point Likert Scale covering the following domains; usefulness, ease of use, ease of learning, satisfaction and intention to use
Investigator feedback | From date of enrollment until end of study completion (24 hours)
  Global impression score

CONTACTS AND LOCATIONS:
Locations (1):
- Falls and Syncope Service, Older People's Medicine, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Protocol, ICF will be made avalible as supplementary material along with a manscript once the study and data analysis has been completed.
Supporting Information: Study Protocol, ICF, CSR